CLINICAL TRIAL: NCT04830995
Title: Impact of High-Intensity Interval Training on Insulin Resistance During Pregnancy: A Randomized Control Trial.
Brief Title: Insulin Sensitivity Response to High-Intensity Training in Insulin Resistance During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Heba mohamed Embaby (Unknown); Salwa Elgendy (Unknown)
Responsible Party: Principal Investigator, Ghada Ebrahim El Refaye, assistant professor Department of Physical Therapy for Women's Health, Faculty of Physical therapy, Cairo University, Egypt, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cairo Un100
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: High Intensity Interval Training; Diet, Healthy
Keywords: Training; Insulin Resistance; Pregnancy
MeSH Terms: conditions — Insulin Resistance | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: group (A) received HIIT and low diet for four weeks, 3 sessions weekly. While the control group received diet only.
Who Masked: Participant, Investigator
Masking Description: Randomization was done by sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diet program (Experimental): moderate restricted diet (1800-2000 kcal/day) for four weeks, 3 sessions weekly
  Interventions: Dietary Supplement: moderate restricted diet (1800-2000 kcal/day) for four weeks
- high intensity interval training (Experimental): high intensity interval training for four weeks, 3 sessions weekly
  Interventions: Dietary Supplement: moderate restricted diet (1800-2000 kcal/day) for four weeks

INTERVENTIONS:
Dietary Supplement: moderate restricted diet (1800-2000 kcal/day) for four weeks — high intensity interval training 3 sessions for four weeks
  Other Names: high intensity interval training

SUMMARY:
Insulin Resistance is one of the common complications that occur during pregnancy. Early intervention is essential to prevent the development of the diseaseThere is evidence that physical inactivity increases the risk of a lot of adverse health problems, including coronary heart disease, type 2 diabetes, breast and colon cancers. It also shortens life expectancy. Pregnancy is a period in the life of women that is often associated with decreased daily physical activity and decreased participation in sports and exercise . In the first few weeks of pregnancy, maternal carbohydrate metabolism is affected by a rise in maternal levels of estrogen and progesterone that stimulates pancreatic β-cell hyperplasia and insulin secretion. As pregnancy progress, pancreatic islet cell hypertrophy continues and there is an increased insulin response to glucose or meal stimulation.

DETAILED DESCRIPTION:
This study was carried out upon twenty multigravida pregnant female between 5-6 months gestation with IR calculated by HOMA test (fasting blood glucose× fasting insulin) ÷ 22.5. Fasting blood glucose was assessed by the method approved by (7, 13) .The test materials for this method were supplied as kits by "Diamond Diagnostics," while Insulin concentrations were stated in formerly frozen and defrosted serum samples by enzyme immunoassay using the human Insulin ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* forty multigravida females.
* their age ranged between 25 to 35 years old.
* Body mass index (BMI) <30kg/ m².

Exclusion Criteria:

* females with pelvic pathology as endometriosis.
* females have irregular menstrual cycles.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-24 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Fasting blood glucose level | three months
  Fasting blood glucose level were measured by expert specialist before and after intervention period from 24th to 37th weeks of pregnancy.

SECONDARY OUTCOMES:
Fasting Insulin Level | three months
  Fasting blood insulin level were measured by expert specialist before and after intervention period from 24th to 37th weeks of pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghada Elrefaye, Giza, Egypt